CLINICAL TRIAL: NCT07034937
Title: Effect of Combination Aerobic and Resistance Training on Diaphragm Excursion Value and Pulmonary Functions in Post Coronary Artery Bypass Grafting Patients
Brief Title: Aerobic and Resistance Training in Post-CABG Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Dr. Hasan Sadikin General Hospital, Bandung, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKFR-202506.01
Record Dates: First submitted 2025-06-09; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Post Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Artery Disease | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Single Group Assignment (Pretest-Posttest)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic and Resistance Training Group (Experimental)
  Interventions: Other: Combination of aerobic training (treadmill walking) and resistance training

INTERVENTIONS:
Other: Combination of aerobic training (treadmill walking) and resistance training — Combination of aerobic training (treadmill walking) and resistance training using resistance bands for deltoid, biceps, triceps, and quadriceps muscles. Conducted twice weekly for 6 weeks (12 sessions). Tools include treadmill and theraband loop bands.

SUMMARY:
This study investigates the effect of combined aerobic and resistance training using resistance bands on diaphragmatic excursion and pulmonary function (FVC, FEV₁, PEF) in post-CABG patients undergoing phase II cardiac rehabilitation.

DETAILED DESCRIPTION:
This quasi-experimental study with a pretest-posttest design evaluates the impact of a 6-week structured aerobic and resistance training program using resistance bands on the diaphragm excursion and pulmonary function. Conducted at the rehabilitation polyclinics of Hasan Sadikin and Al Ihsan hospitals, this study includes post-CABG patients meeting specific inclusion criteria. Intervention is performed twice a week and includes treadmill walking and upper/lower limb resistance exercises. Outcomes will be assessed via ultrasound for diaphragm excursion and spirometry for lung function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients post-CABG surgery maximum 12 weeks after the procedure
2. Age 40-65 years
3. Visual and hearing health
4. Ready to participate in research and sign informed consent.

Exclusion Criteria:

1. Blood pressure greater than 160 mmHg for systolic and diastolic blood pressure greater than 100 mmHg
2. Patients with contraindications to aerobic and resistance training, such as fractures that limit movement.
3. Patients undergoing other therapies that may affect diaphragmatic muscle measurement results, such as electrical diaphragmatic stimulation.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Diaphragm Excursion (cm) | Baseline to Week 6
  The vertical movement of the diaphragm during the respiratory cycle shows the function and mobility of the diaphragm in the process of pulmonary ventilation. The data obtained is expressed in cm.
  Measured via ultrasound.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline to Week 6
  Lung function Forced Vital Capacity (FVC) is commonly assessed through spirometry and measured in liters (L) FVC: This measures the total volume of air that can be forcibly exhaled after a full inhalation. FVC values less than 80% of the predicted value are indicative of restrictive respiratory impairments, where the lungs cannot fully expand. FVC values equal to or greater than 80% are considered normal.
Forced Expiratory Volume in one second (FEV1) | Baseline to Week 6
  Lung function Forced Expiratory Volume in one second (FEV1) is commonly assessed through spirometry and measured in liters (L) FEV1: This represents the air volume a person can forcefully exhale in the first second of a breath.
Peak Expiratory Flow (PEF) | Baseline to Week 6
  Peak Expiratory Flow (PEF) is a spirometric parameter that measures the maximum airflow achieved at the beginning of a forced expiration, expressed in liters per second or minute. It reflects the function of the large airways and expiratory muscle strength. PEF interpretation is based on the percentage of predicted values according to age, sex, and height: ≥80% is considered normal, 60-79% indicates a mild reduction, 40-59% moderate reduction, and <40% signifies a severe reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Dian M Sari, MD., M.Sc., Ph.D, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung

IPD SHARING:
Plan to Share IPD: No